CLINICAL TRIAL: NCT02070653
Title: Does Ticagrelor Inhibit Growth of Small Abdominal Aortic Aneurysms? A Randomised Controlled Trial (TicAAA)
Brief Title: The Efficacy of Ticagrelor on Abdominal Aortic Aneurysm (AAA) Expansion
Acronym: TicAAA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UpAAA - 2014 - 01
Record Dates: First submitted 2014-02-21; First posted 2014-02-25 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-05

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: Aorta; Aneurysm; Antiplatelet
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Aneurysm | interventions — Ticagrelor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ticagrelor (Active Comparator): Ticagrelor 90 mg tablets twice daily for 12 months.
  Interventions: Drug: Ticagrelor
- Placebo (Placebo Comparator): Ticagrelor-placebo tablets twice daily for 12 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ticagrelor
  Arms: Ticagrelor
Drug: Placebo
  Arms: Placebo

SUMMARY:
Abdominal aortic aneurysm (AAA) is a major health problem and ruptured AAA is a common cause of death in Europe and North America. A key limitation of contemporary treatment strategies of AAA is the lack of therapy directed at reducing expansion. Although surgical repair is an effective treatment for large AAA, it is associated with significant mortality and morbidity as well as substantial cost. The rationale for this randomized controlled study is to investigate whether treatment with Ticagrelor inhibits growth of small abdominal aortic aneurysms.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Male and female patients
* Age 50-85 years
* Documented infrarenal aortic aneurysm between 35-49 mm
* Acetylsalicylic acid (ASA)-naïve

Exclusion Criteria:

* Short expected survival.
* On anti-platelet therapy.
* On long-term oral or parenteral anticoagulant treatment.
* On strong inhibitors of CYP3A enzyme (Ketoconazole, Itraconazole, Voriconazole, Telithromycin, Clarithromycin, Ritonavir, Saquinavir, Nelfinavir, Indinavir, Atazanavir).
* On CYP3A (Cytochrome P450, family 3, subfamily A) substrates or inducers >40mg daily doses (Simvastatin, Lovastatin, Rifampin/rifampicin, Phenytoin, Carbamazepine, Phenobarbital).
* Known or suspected connective tissue disorder (Marfans syndrome, etc), infected or inflammatory aneurysm, aneurysm post aortic dissection or previous surgery of the infrarenal aorta.
* Increased risk for bradycardia or ongoing treatment with any bradycardia inducing drug.
* Contraindication for Ticagrelor; hypersensitivity to Ticagrelor or any of the excipients, active pathological bleeding, history of intracranial hemorrhage, moderate or severe hepatic impairment (eg, ascites and/or clinical signs of coagulopathy), on haemodialysis.
* Known haemostatic or coagulation disorder, gastrointestinal bleeding within the past 6 months, or increased bleeding risk due to surgery or trauma within 30 days.
* MRI exclusion criteria, such as: severe claustrophobia, pacemaker, metallic implants in brain, cochlear implants.
* Metallic implants in aortic region.
* Enrolled in either another investigational drug or medical device study or another investigational study of an approved drug or medical device within 30 days prior to visit 1 of the current study.
* Any condition or laboratory finding which in the opinion of the Investigator makes the patient unsuitable for inclusion (eg, active malignancy other than squamous cell or basal cell skin cancer, long-term concomitant treatment with non-steroidal anti-inflammatory drugs (NSAIDs).

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
AAA volume growth | 12 months
  To determine mean reduction in AAA volume growth rate (%) measured with magnetic resonance imaging (MRI) at 12 months

SECONDARY OUTCOMES:
AAA diameter growth, need for surgery and rupture | 12 months
  To determine mean reduction in diameter growth rate (mm), measured with MRI and ultra sound (US), mean reduction in thrombus volume enlargement rate (%) measured with MRI, need for surgery (≥55mm), aneurysm rupture, at 12 months

OTHER OUTCOMES:
Bleeding | 12 months
  To determine bleeding events; primary according to BARC (Bleeding Academic Research Consortium) and secondary according to TIMI (Thrombolysis in Myocardial Infarction) Major and Minor.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Wanhainen, MD. PhD, Principal Investigator — Uppsala University, Sweden
Locations (1):
- Department of Surgical Sciences/Vascular Surgery, Uppsala University, Uppsala, Sweden

REFERENCES:
- [Derived] Wanhainen A, Mani K, Kullberg J, Svensjo S, Bersztel A, Karlsson L, Holst J, Gottsater A, Linne A, Gillgren P, Langenskiold M, Hultgren R, Roy J, Gilgen NP, Ahlstrom H, Lederle FA, Bjorck M. The effect of ticagrelor on growth of small abdominal aortic aneurysms-a randomized controlled trial. Cardiovasc Res. 2020 Feb 1;116(2):450-456. doi: 10.1093/cvr/cvz133. PMID 31135888